CLINICAL TRIAL: NCT04836130
Title: Evaluation of The Accuracy of Zygomatico- Maxillary Complex (ZMC) Fractures Reduction Using Patient Specific Guide (PSG) Versus Conventional Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed Morad (Other)
Responsible Party: Sponsor-Investigator, Ahmed Morad, lecturer assistant, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Omfs 3.3.10
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Zygomatic Fractures
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (ZMC) Fractures reduction Using Patient Specific Guide (PSG) (Active Comparator)
  Interventions: Procedure: patient specific guide
- (ZMC) Fractures reduction Using Conventional Technique (Active Comparator)
  Interventions: Procedure: conventional technique

INTERVENTIONS:
Procedure: patient specific guide — patient specific guide reduction
  Arms: (ZMC) Fractures reduction Using Patient Specific Guide (PSG)
Procedure: conventional technique — conventional anatomical reduction
  Arms: (ZMC) Fractures reduction Using Conventional Technique

SUMMARY:
Evaluation of The Accuracy of Zygomatico- Maxillary Complex (ZMC) Fractures reduction Using Patient Specific Guide (PSG) Versus Conventional Technique

ELIGIBILITY:
Inclusion Criteria:

* • Zygomatic Fracture Type III, IV and V according to rowe and killey classification(13)

  * Age (18-60 years)
  * Recent fracture (less than 2 weeks)

Exclusion Criteria:

* • Zygomatic Fracture Type I, II and VI according to rowe and killey classification(13)

  * Medical compromised patient
  * Patient on radiotherapy
  * Bone disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
accuracy of reduction of the fractured zygoma ( facial asymetry ) | up to 6 months
  assessed by ct

SECONDARY OUTCOMES:
operation time | up to 6 months
  in hours

IPD SHARING:
Plan to Share IPD: Undecided